CLINICAL TRIAL: NCT03279211
Title: True Ileal Amino Acid Digestibility of Whey and Zein Proteins in Healthy Volunteers With Naso-ileal Tubes
Brief Title: Amino Acid Digestibility of Whey and Zein Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, Clinical Head of Gastroenterology, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PROTEOS
Record Dates: First submitted 2017-07-18; First posted 2017-09-12 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Amino Acid
Keywords: digestibility; whey protein; zein; bioavailability

STUDY DESIGN:
Intervention Model Description: 3 groups, one for each protein sources (zein and whey) and one for determination of endogenous amino acid losses (protein-free meal)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zein protein (Experimental): Zein protein included in the test-meal, 30 g of zein in 500 ml (water + flavour/sugar)
  Interventions: Other: Zein Sigma-Aldrich W555025
- Whey protein isolate (Experimental): Whey protein isolate included in the test-meal, 30 g of zein in 500 ml (water + flavour/sugar)
  Interventions: Other: Whey Protein Isolate 894 Fonterra
- Protein-free (Other): No protein added in the test-meal, only 500 ml of water + flavour/sugar In order to determine the endogenous loss of amino acid in the digesta samples.
  Interventions: Other: Protein-free test-meal

INTERVENTIONS:
Other: Whey Protein Isolate 894 Fonterra — 30 g of protein powder diluted in water
  Arms: Whey protein isolate
Other: Zein Sigma-Aldrich W555025 — 30 g of protein powder diluted in water
  Arms: Zein protein
Other: Protein-free test-meal — No protein included in the drink made of water and flavour/sugar
  Arms: Protein-free

SUMMARY:
The main goal of the study is to determine true ileal amino acid digestibility of whey protein isolate (WPI) and zein proteins in healthy subjects equipped with naso-ileal tube. The endogenous losses of proteins and amino acids will be determined by collecting digesta samples after a protein-free diet in a third group of subjects.

DETAILED DESCRIPTION:
True ileal amino acid digestibility of whey protein isolate (WPI) and zein proteins will be determined in healthy subjects. The endogenous losses of proteins and amino acids will be determined by collecting digesta samples after a protein-free test-meal in a different group of subjects.

24 volunteers will be included in the study (men and women; aged 18-65 y; BMI 18-30 kg/m2) and tested at AgroParisTech (Human Nutrition Research Centre of Avicenne Hospital). Due to the invasive procedure of intubation, each volunteer will test only one test-meal (n=8 / test-meal).

One week before the experiment, the volunteers will follow a standard diet adapted to their body weight to control their protein intake (1.3 g protein/kg body weight). The volunteers will arrive at the hospital the morning before the day of the experiment and will be equipped with a double lumen intestinal tube that will be allowed to progress through the intestinal tract for 24h. On the day of the experiment, the position of the tube will be checked by radiography to verify its location at the terminal ileum. A catheter will be inserted in the forearm vein for blood sampling. A perfusion of the non-absorbable marker polyethylene glycol -4000 will start to estimate the intestinal flow and the basal ileal sample will be collected during 30 min. Basal plasma sample will be collected. Then, at t=0, the volunteer will drink the test-meal. Until t=9h, intestinal content will be continuously collected by aspiration and pooled every 30 minutes. Blood will be sampled every 30 minutes during 4h and hourly thereafter.

The test meal will consist of a protein-free biscuit (160 g) and a drink (500 ml) with the test protein as the sole source of protein or no protein for the protein-free group. Celite will be added to the protein-free biscuit and inulin labelled with carbon 13 will be added to the drink as indigestible markers of the meal to allow correction for incomplete collection of digesta. The test proteins will be WPI or zein.

The total nitrogen will be measured in meal and digesta samples by the coupling of Elemental Analysis with stable Isotope Ratio Mass Spectrometry (EA-IRMS) and the amino acid concentration in meal, digesta and plasma samples will be measured by High Performance Liquid Chromatography (HPLC) in order to determine the ileal bioavailability of amino acid of zein and whey protein. Plasma hormonal profile will also be determined to evaluate the effect of each protein sources on metabolic hormones such as insulin, glucagon, leptin, etc.

ELIGIBILITY:
Inclusion Criteria:

* Normal body weight (18 < BMI < 30 kg.m-2)
* Women or men
* 18 - 65 y
* Healthy
* Insured under the French social security system
* Signed informed consent
* For women: use of birth control

Exclusion Criteria:

* People under trusteeship
* Latex, cow milk or corn allergy A
* HIV, hepatite C virus antibodies, hepatite B virus surface antigen and core antibodies positive
* Pregnant women
* Excessive alcohol drinking or drugs intake
* Hypertension, diabetes, digestive tract, liver or renal diseases, severe heart disease
* High sport practicing (> 7h/week)
* Blood donation in the 3 months prior to the study
* Participation in a clinical study in the 3 months prior to the study
* No signed informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Determination of the concentration of amino acids from dietary sources (whey or zein) in the ileal digesta collected during 9 hours after meal intake to calculate the digestibility of amino acids from whey or zein protein sources. | Hour 0 to 9 after intake
  The quantity of amino acids will be determined by HPLC in the ileal digesta collected thanks to the naso-ileal tube during 9 hours after the meal intake. The obligatory endogenous amino acid losses will be estimated by determination of the amino acid content of ileal digesta after intake of the protein-free meal and this value will be subtracted to the values obtained after intake of protein meal to evaluate the quantity of amino acid which comes from dietary sources. Recovery of the indigestible markers (13C-inulin and celite) will allow correction for incomplete collection of digesta.

SECONDARY OUTCOMES:
Determination of the metabolic hormones plasma profile after zein or whey protein intake | Hour 0 to 9 after intake
  Blood will be collected hourly during the 9 hours following the intake of the meal containing zein or whey protein. The profile of concentration of metabolic hormones (amylin, C-peptide, ghrelin, gastric inhibitory polypeptide, glucagon-like peptide 1, glucagon, interleukin -6, insulin, leptin, pancreatic polypeptide, polypeptide tyrosine tyrosine , tumor necrosis factor -α) in plasma will be determined by multiplex hormones assays kit.
Determination of the effect of zein and whey protein on glucose homeostasis | From the evening before the administration to 9 h after the meal.
  Subjects are administered oral deuterated water the day before the investigation. Gluconeogenesis is assessed by measuring deuterium enrichment in body water and on C5 glucose position.
Determination of the effect of zein and whey protein on amino acid plasma concentration | From the evening before the administration to 9 h after the meal.
  Blood will be collected hourly during the 9 hours following the intake of the meal containing zein or whey protein. The profile of concentration of amino acids in plasma will be determined by ultra high performance liquid chromatography.

CONTACTS AND LOCATIONS:
Locations (1):
- CRNH Ile de France, Bobigny, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calvez J, Benoit S, Piedcoq J, Khodorova N, Azzout-Marniche D, Tome D, Benamouzig R, Airinei G, Gaudichon C. Very low ileal nitrogen and amino acid digestibility of zein compared to whey protein isolate in healthy volunteers. Am J Clin Nutr. 2021 Jan 4;113(1):70-82. doi: 10.1093/ajcn/nqaa274. PMID 33021640